CLINICAL TRIAL: NCT03647722
Title: Assessing the Induction of Long-term Immune Regulation Following Treatment With Lemtrada® (Alemtuzumab).
Status: Terminated | Type: Observational
Why Stopped: Study funding was terminated.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Brett T. Lund, Assistant Professor, Neurology, University of Southern California
Other Study IDs: LemRegUSC
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Lemtrada treated - 6 month: Patients that received their first course of treatment with Lemtrada approximately 6 months prior.
  Interventions: Other: Assessment of leukocyte function.
- Lemtrada treated - 12 month: Patients that received their first course of treatment with Lemtrada approximately 12 months prior but who have not received the second course of treatment.
  Interventions: Other: Assessment of leukocyte function.
- Lemtrada treated - 18 month: Patients that received their first course of treatment with Lemtrada approximately 18 months prior and their second course of treatment with Lemtrada approximately 6 months prior.
  Interventions: Other: Assessment of leukocyte function.
- Lemtrada treated - 24 month: Patients that received their first course of treatment with Lemtrada approximately 24 months prior and their second course of treatment with Lemtrada approximately 18 months prior and who have not received any further treatment.
  Interventions: Other: Assessment of leukocyte function.
- Lemtrada qualified - untreated: Patients that are qualified to start treatment with Lemtrada but have not yet being untreated.
  Interventions: Other: Assessment of leukocyte function.

INTERVENTIONS:
Other: Assessment of leukocyte function. — The function and phenotype of regulatory B-cells, regulatory T-cells and alternatively-activated monocytes will be assessed directly ex vivo from PBMC.

SUMMARY:
In this study the investigators wish to test the hypothesis that treatment with Lemtrada is associated with alterations in immune homeostasis in favor of multiple regulatory leukocyte populations which persist long after completion of the treatment phase. Specifically, the investigators propose that regulatory B-cells are induced rapidly following the first course of treatment with Lemtrada, that this occurs prior to induction of other regulatory populations, and that these cells are functionally capable of regulating immune responses. The investigators also propose that there is a concomitant induction of functional regulatory T-cells and alternatively-activated monocytes during the first year after treatment giving a "blanket" enhanced regulatory immune profile. This study is designed primarily to identify possible mechanisms by which Lemtrada acts to modify the immune environment in recipient patients, as such the "outcome" measures are all immunological.

ELIGIBILITY:
Inclusion Criteria:

* Patient must qualify to receive treatment with Lemtrada according to the USC, Department of Neurology, MS Group Clinical Lemtrada Protocol.
* Patient must have been diagnosed with clinically definite Multiple Sclerosis defined by the revised McDonald criteria (Polman et al., 2005, Polman et al., 2010) of the relapsing-remitting form with an Expanded Disability Status Scale (EDSS) score of 0 to 5.5.
* Patient must have the ability to understand and sign this study-specific IRB-approved informed consent form.
* Patients must be willing to donate 80mls of blood for immunological testing either prior to receiving Lemtrada or 6, 12, 18 or 24 months after first round of treatment.

Exclusion Criteria:

* Patient does not qualify to receive treatment with Lemtrada according to the USC, Department of Neurology, MS Group Clinical Lemtrada Protocol.
* Inability to understand nature of the study.
* Patient has any form of progressive MS.
* Patient has been diagnosed with any other autoimmune disease.
* Patient is of child bearing age with a positive pregnancy test or is unwilling to agree to use a reliable contraceptive method.
* Treatment with any of the following within 30 days of commencing treatment with Lemtrada or collection of baseline blood sample: Gilenya, Aubagio, Tecfidera.
* Treatment with Natalizumab within 60 days of commencing treatment with Lemtrada or collection of baseline blood sample.
* Treatment with any of the following within 6 months of commencing treatment with Lemtrada or collection of baseline blood sample: Rituximab, Ocrevus.
* Treatment at any time with any of the following: Mitoxantrone, Cyclophosphamide, Cladribine, Cyclosporine, Azathioprine, Methotrexate or any other immunomodulatory, immunosuppressant or immune homeostasis altering drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit 125 individuals with clinically definite MS, defined by the revised McDonald criteria (35). Patients in each cohort will be enrolled from those currently being seen by physicians at the University of Southern California, Department of Neurology.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Assess changes in the circulating regulatory B-cell population. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Brett T Lund, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Department of Neurology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kashani N, Kelland EE, Vajdi B, Anderson LM, Gilmore W, Lund BT. Immune Regulatory Cell Bias Following Alemtuzumab Treatment in Relapsing-Remitting Multiple Sclerosis. Front Immunol. 2021 Oct 28;12:706278. doi: 10.3389/fimmu.2021.706278. eCollection 2021. PMID 34777337